CLINICAL TRIAL: NCT02018367
Title: Accuracy, Yield and Clinical Impact of a Low-Cost High Resolution Microendoscope in the Early Diagnosis of Esophageal Adenocarcinoma
Brief Title: Accuracy, Yield and Clinical Impact of a Low-Cost HRME in the Early Diagnosis of Esophageal Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Collaborators: William Marsh Rice University (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GCO #12-0289, H-36538
Record Dates: First submitted 2013-12-09; First posted 2013-12-23 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus; proflavine; Microscopic imaging
MeSH Terms: conditions — Barrett Esophagus | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proflavine, high resolution imaging (Experimental): Proflavine hemisulfate will be used as a topical contrast agent in conjunction with the high resolution imaging device to visualize and image areas suspicious for neoplasia. Biopsies will be taken per Seattle biopsy protocol for Barrett's Esophagus surveillance.
  Interventions: Drug: Proflavine, high resolution imaging
- Standard of care (No Intervention): Standard of care examination of the upper GI tract using the standard high resolution endoscope with bipsies taken per Seattle biopsy protocol for Barrett's Esophagus surveillance.

INTERVENTIONS:
Drug: Proflavine, high resolution imaging — 5-10mL of proflavine hemisulfate (0.01%) will be sprayed on the esophageal mucosa. The HRME will then be inserted through the biopsy channel of the endoscope and gently placed against the mucosa. The endoscopist will image each discrete lesion observed during white light endoscopy. For each HRME imaged area, an optical read will be obtained followed by a tissue biopsy.
  Other Names: Proflavine hemisulfate
  Arms: Proflavine, high resolution imaging

SUMMARY:
The overall goal of the study is to determine whether imaging with the low-cost High Resolution Microendoscope(HRME) will increase the efficiency and yield of the current standard of endoscopic surveillance of Barrett's esophagus. We believe the HRME will provide an in-vivo "optical biopsy" that will be comparable to gold standard histopathology and allow the endoscopist to make a more informed decision about whether to obtain a biopsy or even perform endoscopic therapy (i.e. endoscopic mucosal resection, EMR).

DETAILED DESCRIPTION:
Primary outcomes:

* the diagnostic yield (defined as the proportion of mucosal biopsy samples with neoplasia) of HRME with directed biopsy

  - compared to standard white-light endoscopy with 4-quadrant random biopsy (WL) for the diagnosis of BE-associated neoplasia in flat mucosa as well as mucosal lesions
* the clinical impact of HRME on the diagnosis and endoscopic surveillance of BE- associated neoplasia

  * does HRME alter the decision to obtain a mucosal biopsy or perform endoscopic mucosal resection (EMR)
  * the total number of total mucosal biopsies taken per procedure; does HRME alter the number of biopsies necessary?

Secondary outcomes:

* sensitivity, specificity, positive predictive value, and negative predictive value of HRME for the in-vivo diagnosis of neoplasia in a routine surveillance population of patients with BE (using histopathologic diagnosis of mucosal biopsies as the reference standard)
* the total procedure time for imaging and mucosal biopsy acquisition of HRME - compared with WL, stratified by length of BE (< 3 cm and > 3cm)

ELIGIBILITY:
Inclusion Criteria:

* outpatients with > 1 cm biopsy-proven Barrett's Esophagus who are undergoing standard of care endoscopic surveillance for metaplasia, dysplasia, or neoplasia.

Exclusion Criteria:

* Allergy or prior reaction to the fluorescent contrast agent proflavine
* Patients who are unable to give informed consent.
* Known advanced adenocarcinoma of the distal esophagus, or dysplastic/suspected malignant esophageal lesion > 2 cm in size not amenable to EMR
* Patients with a history of a severe allergic reaction (anaphylaxis)
* Patients unable to undergo routine endoscopy with biopsy :
* Women who are pregnant or breastfeeding
* Prothrombin Time > 50% of control; PTT > 50 sec, or INR > 2.0)
* Inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other
* Patients with known, untreated esophageal strictures, prior partial esophageal resection, or altered anatomy preventing passage of the endomicroscope
* Patients with known severe esophagitis
* Patients with suspected but no biopsy confirmed BE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic yield (defined as the proportion of mucosal biopsy samples with neoplasia) of HRME with directed biopsy | 1 day
  Compared to standard white-light endoscopy with 4-quadrant random biopsy (WL) for the diagnosis of BE-associated neoplasia in flat mucosa as well as mucosal lesions

SECONDARY OUTCOMES:
The diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of HRME for the in-vivo diagnosis of neoplasia. | 1 day
  To be determined using histopathologic diagnosis of mucosal biopsise as the reference standard

OTHER OUTCOMES:
The clinical impact of HRME on the diagnosis and endoscopic surveillance of BE- associated neoplasia | 1 day
  Does HRME alter the decision to obtain a mucosal biopsy or perform endoscopic mucosal resection (EMR) The total number of total mucosal biopsies taken per procedure; does HRME alter the number of biopsies necessary?

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Anandasabapathy, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Shin D, Lee MH, Polydorides AD, Pierce MC, Vila PM, Parikh ND, Rosen DG, Anandasabapathy S, Richards-Kortum RR. Quantitative analysis of high-resolution microendoscopic images for diagnosis of neoplasia in patients with Barrett's esophagus. Gastrointest Endosc. 2016 Jan;83(1):107-14. doi: 10.1016/j.gie.2015.06.045. Epub 2015 Aug 5. PMID 26253018

DOCUMENTS (3):
  • Informed Consent Form (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02018367/ICF_000.pdf
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02018367/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02018367/SAP_002.pdf